CLINICAL TRIAL: NCT06414213
Title: Enhancing Locomotor Learning With Motor Imagery and Transcranial Direct Current Stimulation
Brief Title: Improving Locomotor Learning With Brain Stimulation
Acronym: ELLMITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Principal Investigator, Jared W Skinner, Assistant Professor, Appalachian State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-21-0198
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Motor Learning
Keywords: randomized; double-blinded; tDCS; motor imagery; functional near-infrared spectroscopy (fNIRS); controlled trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- MI/Active tDCS (Experimental): The participants received active tDCS current and participated in the Motor Imagery intervention.
  Interventions: Behavioral: Motor Imagery (MI); Device: Active tDCS
- MI/Sham tDCS (Sham Comparator): The participants received sham tDCS current and participated in the Motor Imagery intervention.
  Interventions: Behavioral: Motor Imagery (MI); Device: Sham tDCS
- Control (No Intervention): The control group watched an unrelated (non stimulating) video for a duration equal to the MI groups' intervention tasks.

INTERVENTIONS:
Behavioral: Motor Imagery (MI) — Participants watched a standardized video sequence that consisted of an individual completing twenty walking trials (twenty video clips-each clip represents one trial). Participants were instructed to place their focus intently on the person performing the obstacle course and try to imagine themselves doing the skill. Periodically, a reminder would appear to help focus and redirect participant's attention to different aspects of the video or different versions of imagery (visual or kinesthetic). Participants will watch the video first at normal play speed and then in slow motion after a short break (30 secs to 1 min). Total training time will be approximately 20 mins which is consistent with the duration of the locomotor intervention and duration of stimulation.
  Arms: MI/Active tDCS; MI/Sham tDCS
Device: Active tDCS — The participants received a 20-minute "active" session of tDCS at a 2-milliamp current.
  Arms: MI/Active tDCS
Device: Sham tDCS — The participants received a 20-minute session of "sham" tDCS.
  Arms: MI/Sham tDCS

SUMMARY:
The primary goal of this research was to assess the practicality and initial effectiveness of a motor imagery (MI) intervention combined with elements of action observation (AO), alongside active or sham transcranial direct current stimulation (tDCS) over the prefrontal cortex (PFC), on locomotor learning in healthy adults. Feasibility was determined by examining recruitment rates, participant engagement, and safety measures. The efficacy of the intervention was gauged by analyzing the time taken to complete tasks and changes in cerebral blood flow immediately after the intervention and one week later. The study was guided by three main hypotheses: (1) the intervention techniques would be well-received and safe for the participants; (2) compared to a control group, MI training would lead to better learning outcomes and retention of learning; (3) in comparison to the control and sham tDCS groups, active tDCS would result in superior learning outcomes and retention of learning.

DETAILED DESCRIPTION:
The study implemented a double-blind, randomized, controlled trial design. Participants were tested three times over 7 days. After study enrollment, the participants were randomly assigned to one of three groups: MIActive (receiving active tDCS stimulation and participating in MI protocol), MISham (receiving sham tDCS stimulation and participating in MI protocol), and Control (receiving no stimulation and participating in an unrelated video-watching task) by a research member not associated with data collection. Allocation ratio was 1:1:1 and a block randomization approach was employed to maintain an equal distribution of participants across the three groups throughout the study. Study participants and assessors were blinded to assignment of active or sham tDCS. The independent variables were time (pre, post, and retention trials) and group (MIActive, MISham and Control), and the dependent variables were time to completion of a complex obstacle course and the amount of change in oxygenated hemoglobin (ΔO2Hb) during performance of that task.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults age 18 and older
* Freely ambulatory (no assistive walking aids)

Exclusion Criteria:

* Failure to meet specific inclusion criteria
* History or presence of any neurological disease
* Low visual ability, operationally defined as visual acuity less than 20/70 on the standard eye chart
* Extreme difficulty performing walking tasks due to low visual ability
* Clinical judgment of the investigative team
* Additionally, subjects who are determined to be at increased risk for adverse events during the tDCS procedure, as determined by the tDCS screening questionnaire

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared W Skinner, PhD, Principal Investigator — Appalachian State University
Locations (1):
- Appalachian State University, Boone, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make Individual Participant Data (IPD) available.

REFERENCES:
- [Background] Clark DJ, Chatterjee SA, Skinner JW, Lysne PE, Sumonthee C, Wu SS, Cohen RA, Rose DK, Woods AJ. Combining Frontal Transcranial Direct Current Stimulation With Walking Rehabilitation to Enhance Mobility and Executive Function: A Pilot Clinical Trial. Neuromodulation. 2021 Jul;24(5):950-959. doi: 10.1111/ner.13250. Epub 2020 Aug 18. PMID 32808403
- [Derived] Gamwell-Muscarello HE, Needle AR, Meucci M, Skinner JW. Improving locomotor performance with motor imagery and tDCS in young adults. Sci Rep. 2025 Jan 11;15(1):1748. doi: 10.1038/s41598-025-86039-2. PMID 39799141

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control
Started | 13 | 12 | 13
Completed | 12 | 11 | 10
Not Completed | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: participants were excluded if they did not attend the follow up session
Groups:
- Total: Total of all reporting groups
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control | Total
Number analyzed (Participants) | 13 | 12 | 13 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 13 | 38
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.42 (1.98) | 22.36 (2.06) | 24.1 (4.04) | 22.96 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 10 | 32
  Male | 2 | 1 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Prefrontal Cortical Activity
Description: Functional near infrared spectroscopy (fNIRS) monitor (OctaMon by Artinis Medical Systems), changes in oxygenated hemoglobin concentration (O2Hb) relative to a baseline task
Time Frame: Baseline to 1 week follow up
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control
Number analyzed (Participants) | 12 | 11 | 10
μM
  Baseline (Pre-Intervention) | 0.04 (0.47) | 0.11 (0.68) | 0.58 (0.50)
  20 minutes post Baseline (Post-Intervention) | -0.62 (0.70) | -0.19 (0.91) | 0.20 (0.81)
  1 Week Follow up | -0.61 (0.51) | 0.24 (1.11) | 0.12 (0.64)

2. Primary Outcome: Adherence to Interventions
Description: number of sessions attended
Time Frame: Baseline to 1 week follow up
Measure: Mean (Standard Deviation); unit: Numbers of session completed
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control
Number analyzed (Participants) | 13 | 12 | 13
Numbers of session completed | 1.92 (0.27) | 1.91 (0.28) | 1.77 (.43)

3. Primary Outcome: Retention of Participants
Description: number of participants completing intervention and follow-up assessment
Time Frame: Baseline to 1 week follow up
Measure: Count of Participants; unit: Participants
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control
Number analyzed (Participants) | 13 | 12 | 13
Participants | 12 | 11 | 10

4. Primary Outcome: Adverse Events in Each Study Arm
Description: Number of unexpected and/or serious adverse events
Time Frame: Baseline to 1 week follow up
Measure: Number; unit: number of adverse events
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control
Number analyzed (Participants) | 12 | 11 | 10
number of adverse events | 0 | 0 | 0

5. Primary Outcome: Time to Completion
Description: Recorded time to complete the obstacle course
Time Frame: Baseline to 1 week follow up
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control
Number analyzed (Participants) | 12 | 11 | 10
seconds
  Baseline/Pre | 46.60 (7.8) | 47.64 (6.42) | 39.27 (8.1)
  Post-Test | 40.72 (3.45) | 47.21 (4.3) | 37.2 (7.8)
  1 Week Follow up | 39.1 (3.98) | 45.43 (3.8) | 36.1 (8.3)

6. Secondary Outcome: Kinesthetic and Visual Imagery Questionnaire (KVIQ)
Description: The Kinesthetic and Visual Imagery Questionnaire (KVIQ-10) measures the ability to imagine movements. This test evaluates the subject's ability to see (visual imagery) and feel (kinesthetic imagery) movements. The KVIQ-10 total score ranges from 10 to 50 (visual and kinesthetic subscale scores each range from 5 to 25).The KVIQ consists of 10 items, (5 movements for each scale), each item being a separate movement followed by rating the ease or difficulty of generating those self-images on a 5-point Likert scale (where 1 = no image or sensation and 5 = Image as clear as seeing or as intense as executing the action). Higher scores reflect higher imagery abilities.
Time Frame: Baseline to 1 week follow up
Population: The motor imagery/active tDCS and motor imagery/sham tDCS groups participated in the KVIQ-10 assessments, receiving motor imagery and active or sham transcranial direct current stimulation, respectively. These assessments evaluated their kinesthetic and visual imagery abilities, in order to compare their relative capabilities. The control group did not participate in the KVIQ-10 because they did not engage in motor imagery training, making the administration of the KVIQ-10 irrelevant for them.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MI/Active tDCS | MI/Sham tDCS
Number analyzed (Participants) | 12 | 11
score on a scale
  External Imagery | 21.3 (4.1) | 22.7 (3.0)
  Kinesthetic Imagery | 22.9 (4.7) | 21.7 (4.5)

ADVERSE EVENTS:
Time Frame: from baseline to follow-up
Arm/Group | MI/Active tDCS | MI/Sham tDCS | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT06414213/Prot_SAP_000.pdf